CLINICAL TRIAL: NCT06269445
Title: The Efficacy and Safety of Lcaritin Combined With Bevacizumab and FOLFIRI in Treatment of Liver Metastases From Colorectal Cancer: A Prospective, Single-arm Study
Brief Title: The Efficacy and Safety of Lcaritin Combined With Bevacizumab and FOLFIRI in Treatment of Liver Metastases From Colorectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Sheng Dai, Principal Investigator, head of medical affairs, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-942-01
Record Dates: First submitted 2024-01-24; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icaritin Combined With Bevacizumab and FOLFIRI (Experimental): Icaritin: 600 mg orally, bid; Bevacizumab: Intravenous infusion, 5 mg/kg per dose, every 14 days; FOLFIRI: ①Irinotecan: Irinotecan should be given on the first day of chemotherapy at a dose of 180mg/m2 by intravenous drip.The infusion time should be >30-90min.
  ②Calcium folinate: give irinotecan at a dose of 400mg/m2 by intravenous drip in conjunction with irinotecan infusion, and the infusion time should be up to 2h.
  ③5-fluorouracil: give intravenous infusion at a dose of 400mg/m2 on the first day of chemotherapy, then give an intravenous drip at a dose of 1200mg/m2 for 2 days, the total amount of 2400mg/m2 , and continue to be infused for 46-48h.
  Interventions: Drug: Icaritin Combined With Bevacizumab and FOLFIRI

INTERVENTIONS:
Drug: Icaritin Combined With Bevacizumab and FOLFIRI — Bevacizumab and FOLFIRI are second-line treatment options for colorectal cancer; synergistic efficacy expected in combination with Icaritin

SUMMARY:
To evaluate the efficacy and safety of the combination regimen of Icaritin with bevacizumab + FOLFIRI in patients with liver metastases from advanced colorectal cancer.

DETAILED DESCRIPTION:
At present, second-line only targeting combined with chemotherapy is the main treatment option, and the choice of treatment modality is limited, with the immunotherapy rise of immunotherapy, the mode of combining immunotherapy on the basis of existing first- and second-line chemotherapy combined with targeting is also being actively explored, but no positive results of large-scale phase III clinical studies have been reported yet. Meanwhile, there is no solution to the the problem of pro-inflammatory factor release. Therefore, it is necessary to consider the combination of a drug with a better safety profile and target-immunity synergistic effect. A combination of drugs with better safety and target-immunity synergistic effect could be considered as a safer and more effective treatment option for patients with liver metastases from advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1). Age ≥ 18 years. 2).Patients with unresectable advanced metastatic colorectal cancer confirmed by clinical diagnostic criteria and/or histopathological or cytological examination. Metastases include, but are not limited to the liver.

  3). Presence of clearly measurable (RECIST 1.1 compliant) liver metastases on imaging assessment (unresectable by MDT assessment).

  4). Patients who have failed prior first-line systemic systemic therapy, including bevacizumab.

  5).ECOG PS score 0-1. 6). Have normal organ function and meet the following criteria on laboratory tests within 7 days prior to initiation of therapy:
  1. Haemoglobin level > 80 g/L;
  2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
  3. Platelet count ≥50×10-9/L;
  4. Serum albumin ≥ 30 g/L;
  5. Total bilirubin ≤ 2 × upper limit of normal (ULN);
  6. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 5 × ULN;
  7. Alkaline phosphatase (ALP) ≤ 2.5 x ULN;
  8. creatinine ≤ 1.5 x ULN and creatinine clearance ≥ 50 ml/min. 7). Good swallowing function. 8). Coagulation function: international normalised ratio (INR) ≤ 1.5 x ULN or prothrombin time (PT)≤16s.

     9). Life expectancy ˃3 months. 10). Voluntary participation in this study and voluntary signing of informed consent.

     11). Men and women of gestational age must agree to use adequate contraception throughout the study and for 3 months after the end of treatment.

     Exclusion Criteria:
* 1). Pre-existing or coexisting other active malignant tumours (except for malignant tumours that have been curatively treated and have been free of malignancy that has received curative treatment and has been free of morbidity for more than 5 years or carcinoma in situ that can be cured by adequate treatment).

  2). Concomitant administration of modern Chinese medicinal preparations for antitumour and anti-tumour indications.

  3). Patients who have received chemotherapy or anti-vascular endothelial growth factor receptor (VEGF) therapy.

  4). Patients receiving systemic chemotherapy, hormonal therapy, immunotherapy, approved proteins/antibodies or any experimental drugs or treatments (30 days) or radiotherapy (within 14 days).

  5). Tumour invasion of large blood vessels. 6). Significant cardiovascular compromise within 12 months prior to the first dose of study drug: e.g., New York Heart Association (NYHA) Class II or higher. Stroke, myocardial infarction or cerebral haemorrhage, or arrhythmia associated with haemodynamic instability; Corrected QT (QTc) interval prolongation >480ms.

  7). Any surgical procedure within the last 28 days. 8). Bleeding from ruptured oesophageal or gastric varices within the last 2 weeks, or unconfirmed severe varices and bleeding in the judgement of the investigator.

  9). Bleeding or thrombotic disorders or on thrombolytic therapy, coagulation disorders; study intervention Clinically significant haemoptysis or tumour bleeding of any cause within 2 weeks prior to first dose.

  10). Patients with uncontrolled epilepsy, history of central nervous system disease or psychiatric disorders, hypertension.

  11). Active autoimmune disease requiring systemic therapy within the past 2 years.

  12). Clinically significant ascites on physical examination that cannot be controlled medically.

  13). Pregnant or breastfeeding female patients, or those unwilling to use contraception during the trial.

  14). Known hypersensitivity to Icaritin, Bevacizumab and chemotherapeutic drug components.

  15). Suspect that it may cause contraindication to the use of the drug, or affect the reliability of the study results, or place the patient at a disease or condition that places the patient at high risk for treatment complications, or affects the patient's adherence to the trial medication.

  16). Vulnerable populations, including those with mental illness, cognitive impairment, critically ill patients, illiteracy, etc.

  17). Presence of other reasons that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | up to 5 years
  Time between the start of the trial and the onset of (any aspect of) tumour progression or death (from any cause).

SECONDARY OUTCOMES:
Objective remission rate (ORR) | up to 5 years
  The proportion of patients whose tumour volume shrinks to a pre-specified value and who are able to maintain the minimum timeframe requirement is the sum of the proportions in complete and partial remission.
Overall survival (OS) | up to 5 years
  Time from start of trial to death (from any cause).
Disease Control Rate (DCR) | up to 5 years
  Number of cases in remission (PR+CR) and stable lesions (SD) after treatment as a percentage of evaluable cases.
Duration of ongoing remission (DOR) | up to 5 years
  The time from the start of the first assessment of the tumour as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
TRAEs | up to 5 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0
Quality of life of the patients | up to 5 years
  Quality of life of the patients will be assessed by Functional Assessment of Cancer Therapy - Colorectal (FACT-C) questionnaire liscenced from The Functional Assessment of Chronic Illness Therapy System ("FACIT System"). By using the Manual scoring template, some items are reverse scored. Subscale scores, total scores and TOI scores. The higher the score, the better the QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Dai, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The data is expected to be released on Dec 2025, and will be uploaded to http://www.medresman.org.cn/ Clinical Research Data Management Platform
Time Frame: The data is expected to be released on Dec 2025
Access Criteria: Case Record Form